CLINICAL TRIAL: NCT07381036
Title: Comparison of Nebulized Ketamine With Nebulized Magnesium Sulfate for the Prevention of Postoperative Sore Throat in Adult Surgical Patients Undergoing General Anesthesia: Prospective Randomized Controlled Study
Brief Title: Comparison of Nebulized Ketamine With Nebulized Magnesium Sulfate for the Prevention of Postoperative Sore Throat
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shahenda Ahmed Ali, Resident of Anesthesia and surgical Intensive Care unit and Pain Management, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Soh-Med-25-12-7MS
Record Dates: First submitted 2026-01-22; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Sore Throat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketamine group (Experimental)
  Interventions: Drug: Ketamine nebulizer
- Mg sulfate group (Experimental)
  Interventions: Drug: Mg sulfate nebulizer
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine nebulizer — 50 patients will receive preoperative nebulization with 50 mg ketamine in 5 ml normal saline.
  Arms: Ketamine group
Drug: Mg sulfate nebulizer — 50 patients will receive preoperative nebulization with 250 mg magnesium sulfate in 5 ml normal saline.
  Arms: Mg sulfate group
Drug: Placebo — 50 patients will receive preoperative nebulization with 5 ml normal saline.
  Arms: Placebo group

SUMMARY:
The aim of this study is to compare the efficacy of nebulized ketamine versus nebulized magnesium sulfate in reducing the incidence and severity of POST.

* Primary outcome

  • To compare the incidence of POST method.
* Secondary outcomes

  * Onset, Severity, and duration of POST at 0, 2, 4, 6, 12, 24 hours postoperative.
  * The hemodynamics recording (HR, BP, MBP, pre and post nebulization)
  * Adverse Effects (e.g., sedation, cough, nausea, vomiting, ….)

DETAILED DESCRIPTION:
Post-operative sore throat (POST) is a common complication seen in patients after general anesthesia with endotracheal intubation although clinicians often regard it as a minor complication. The incidence of POST is estimated to be 21%-65% in different studies . The primary cause of POST is airway irritation and inflammation or trauma caused by an endotracheal tube; however, the airway may be extremely sensitive due to a preexisting comorbid condition. Regardless of its incidence and some preventive measures, POST is listed from the top as patients' most undesirable outcome in the postoperative period. POST is well recognized that reporting of sore throat is affected by the method of questioning that is whether the questions asked directly or indirectly .

The expression of POST constitutes a number of signs and symptoms. For example, sore throat is an ordinary expression of pharyngitis, which by itself can have a number of causes. It may also include a variety of symptoms including pain and discomfort, laryngitis, tracheitis, hoarseness, cough, or dysphagia. This leads to an increase in morbidity and causes further complications in patients .

Various pharmacological and nonpharmacological methods have been tried to decrease the incidence of POST with varying success rates. The pharmacological methods used for the prevention of POST are the use of inhalational, intravenous or topical agents that include beclomethasone gel, magnesium sulfate gargle, ketamine gargle, nebulized ketamine, magnesium sulfate nebulization, and lidocaine spray .

Nebulized medication administration is strongly recommended over intranasal delivery that is inhaled into the lungs and respiratory tract and is an important strategy for various respiratory problems and diseases. It reduces cough, temporary nasal discomfort, and vocal cord irritation. N-methyl-D-aspartate (NMDA) receptors had a crucial part in inflammation and nociception in the body. NMDA receptors exist in both peripheral nervous system (PNS) neurons and the central NS (CNS) .

Ketamine, an NMDA receptor antagonist, is commonly administered as a nebulizer to decline the severity and frequency of POST owing to its antinociceptive and anti-inflammatory properties .

Magnesium is also another NMDA receptor antagonist that plays a significant role in decreasing the incidence of POST. It is used as nebulizer; it is accessible and easily available in hospitals. The efficacy of preoperative nebulization of magnesium sulfate was assessed and found that the incidence and severity of POST were reduced at rest and on swallowing through 24 hours post extubation (8). Some studies showed that ketamine and magnesium can be used for attenuation of postoperative sore throat .

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Elective surgery requiring GA with endotracheal intubation.

  - Exclusion Criteria:
* Surgery involves the oral cavity, nasopharynx, larynx, and neck regions.
* Surgery requires prone position.
* Surgery lasted more than 3 hours.
* History of preoperative sore throat, common cold.
* Anticipated difficult airway.
* Any known allergies to study drugs.
* Recent non-steroidal anti-inflammatory drugs use.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of Post operative sore throat method. | 24 hours

IPD SHARING:
Plan to Share IPD: Undecided